CLINICAL TRIAL: NCT03227640
Title: The Impact on Ovarian Reserve of Ovarian Cystectomy Versus Laser Vaporization in the Treatment of Ovarian Endometrioma: a Randomized Clinical Trial
Acronym: Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Massimo Candiani, Professor, Scientific Institute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LaserLuM
Record Dates: First submitted 2017-07-09; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Endometrioma
MeSH Terms: conditions — Endometriosis | interventions — Lasers, Gas

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stripping (Active Comparator): standardized laparoscopic stripping technique
  Interventions: Procedure: stripping technique
- CO2 laser vaporization (Experimental): drainage of the cyst content and vaporization of the internal wall with CO2 laser
  Interventions: Device: CO2 laser (AcuPulse Duo, Lumenis)

INTERVENTIONS:
Procedure: stripping technique — The cyst is stripped from the healthy ovary by traction and countertraction; after the removal of the cyst, hemostasis is achieved by selective bipolar coagulation.
  Arms: stripping
Device: CO2 laser (AcuPulse Duo, Lumenis) — The cyst content is drained and the internal wall is vaporized with CO2 laser beam (AcuPulse Duo, Lumenis, Israel)
  Arms: CO2 laser vaporization

SUMMARY:
This is a prospective, multicentric (two centers: 1:San Raffaele Scientific institute, Milan, Italy; 2:Jagiellonian University, Collegium Medicum, Cracow, Poland), randomized (1:1) clinical trial that includes patients undergoing surgery for primary unilateral or bilateral symptomatic endometriomas.

The aim of the study is to determine whether and to what extent the two surgical procedures for endometrioma, cystectomy and laser vaporization, affect ovarian reserve. Recently, cystectomy has been questioned as an ideal surgical approach because it may involve excessive removal of ovarian tissue and the loss of follicles; laser vaporization has been proposed as a promising method to preserve ovarian function.

DETAILED DESCRIPTION:
Excisional surgery is the recommended treatment for ovarian endometrioma because of higher pregnancy rate and lower recurrence rate compared with ablative techniques. From the standpoint of ovarian reserve, the efficiency of cystectomy remains a topic of considerable debate: in recent years, cystectomy has been questioned as an ideal surgical approach for endometriomas because it is associated with excessive removal of ovarian tissue and loss of ovarian follicles with subsequent reduction of ovarian reserve. According to a recent report, absence of follicular growth was observed in 13% of operated ovaries, although this event never occurred in the contralateral gonad.

In San Raffaele Scientific Institute, fear of ovarian failure after cystectomy resulted in the introduction of an ablative technique involving CO2 laser technology, which posses the ability to deliver energy with little thermal spread. More than 80 patients were treated with CO2 laser at this Institution during three-year experience. This surgical procedure was inspired by the one employed by Jacques Donnez for more than 20 years, in which CO2 laser is used to ablate endometriomas' inner wall, after 3-months GnRHa therapy. Laser vaporization, according to the ''three-step procedure", has also been proposed as the best method to preserve ovarian function; moreover, reassuring data on the rate of long-term recurrence after laser vaporization have recently been published.

However, no data are available about the single use of CO2 laser fiber vaporization (without GnRHa therapy) with respect to the ovarian reserve.

Since 2015, the investigators have continuously evaluated the benefits of CO2 laser vaporization through a clinical trial assessing the postoperative changes in ovarian reserve as indicated by antral follicle count (AFC) and anti-mullerian hormone (AMH); the results of this pilot study support the positive effects of CO2 laser on ovarian reserve as demonstrated by higher AFC and no change in AMH at 3-month follow-up. In order to provide more conclusive data about the potential advantage of CO2 laser ablation with respect to ovarian cystectomy in terms of fertility outcomes a prospective randomized trial has been planned; the aim of this prospective randomized study is to determine whether and to what extent the two surgical procedures for ovarian endometrioma (cystectomy versus C02 laser vaporization) affect ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral endometriomas
* pain and/or infertility associated with endometriomas
* largest diameter of the endometrioma ≥3 cm and ≤ 8 cm

Exclusion Criteria:

* intra-operative detection of deep infiltrating endometriosis
* evidence of adenomyosis at the preoperative ultrasound
* previous surgical procedures on the ovaries
* previous unilateral oophorectomy
* previous salpingectomy or hysterectomy
* thyroid disease
* hyperprolactinemia
* diabetes mellitus
* adrenal disorders
* suspected or proven ovarian malignancy
* evidence of premature ovarian failure (POF) or premature menopause
* hormonal treatment within 3 months from baseline ovarian reserve assessment and 3 months after surgery.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-08-01 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
changes in antral follicle count (AFC) | baseline and 3 months
  number of follicles with average diameter of 2-10 mm in both ovaries assessed on the second and fifth day of the menstrual cycle

SECONDARY OUTCOMES:
changes in serum antimullerian hormone (AMH) levels | baseline and 3 months
  AMH is assessed on venous blood samples (Beckman-Coulter 2nd-generation; Gen II) obtained on day 2-5 of the menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Candiani, MD Prof, Principal Investigator — San Raffaele Scientific Institute
Locations (2):
- San Raffaele Scientific Institute, Milan, Italy
- Jagiellonian University, Collegium Medicum, Cracow, Poland, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Candiani M, Ottolina J, Posadzka E, Ferrari S, Castellano LM, Tandoi I, Pagliardini L, Nocun A, Jach R. Assessment of ovarian reserve after cystectomy versus 'one-step' laser vaporization in the treatment of ovarian endometrioma: a small randomized clinical trial. Hum Reprod. 2018 Dec 1;33(12):2205-2211. doi: 10.1093/humrep/dey305. PMID 30299482